CLINICAL TRIAL: NCT05551572
Title: Physiopathology of Prosthetic Joint Infections : a Pilot Study
Brief Title: Physiopathology of Prosthetic Joint Infections
Acronym: PROTHEE-PILOTE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220417
Record Dates: First submitted 2022-06-10; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Prosthetic-joint Infection
Keywords: prosthetic joint infection; prosthesis loosening; Staphylococcus; osteoblast; immune system; microenvironment
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human tissue samples collected during surgery for prosthetic joint infection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- septic samples: patients undergoing revision surgery for prosthetic joint infection
- aseptic samples: patients undergoing revision surgery for prosthetic replacement without infection

SUMMARY:
This study aim to explore cellular responses of bone and immune cells to bacterial infections observed in patients with prosthetic joint infections. The investigators will analyze clinical data and tissue samples collected from patients undergoing surgery as part of their usual care for prosthetic joint infections. These research will be conducted on three different hospitals in Paris: Lariboisière (AP-HP), Cochin (AP-HP) and Croix Saint-Simon.

DETAILED DESCRIPTION:
The number of prosthetic joint infections (PJI) new cases in France is estimated at 2000/2500 cases per year. PJI, mainly caused by staphylococci, are serious infections responsible for significant morbidity result of inflammation and bone destruction (osteomyelitis). Despite optimal medical and surgical management, a risk of failure and recurrence exists, which varies depending on the situation.

In addition to the deterioration in patients' quality of life, the economic cost for the health care system is very high, in particular because of prolonged hospitalizations, complex treatments, and frequent readmissions. Thus, the adequate management of PJI is a major public health issue.

In this context, new therapeutic approaches are urgent medical needs for the management of patients with PJI.

Thus, the identification of the biological mechanisms (immunology, microbiology, bone physiology) underlying these infections is essential. Indeed, the impact of bacterial infections on bone homeostasis is poorly documented. Although several biological mechanisms have been suggested the host-pathogen interaction and the close links between bacterial infection and biological response of bone cells to microorganisms and their environment warrant to be explored.

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old and older
* Patient eligible for lower limb revision surgery (revision surgery for infected or non-infected prosthesis)
* Patient affiliated to a social security system
* Oral consent to the research

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients eligible for lower limb revision surgery for infected or non-infected prosthesis. Primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
markers of bone loss | 12 months
  Immunohistochemistry detection of Tartrate-resistant acid phosphatase cells (TRAP); cathepsin K; Matrix Metalloproteinase 9 (MMP9); sclerostin

SECONDARY OUTCOMES:
markers of cellular activity in the bone microenvironment | 12 months
  immunohistochemistry detection of nuclear factor-activated T cells c1 (NFATc1); Matrix Metalloproteinase 9 (MMP9); Fibroblast growth factor 23 (FGF23)
immune-profiling of bone microenvironment | 12 months
  mapping lymphoid and myeloid cells by spectral flow cytometry assay
inflammatory mediators in the bone microenvironment | 12 months
  flow cytometry quantification of cytokine producing cells
differentiation between osteoclasts from mononuclear phagocytes | 12 months
  enzyme-linked immunosorbent (ELISA) and/or flow cytometry assays using specific antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Martine COHEN-SOLAL, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided